CLINICAL TRIAL: NCT03928873
Title: Extracorporeal Shock Wave Therapy Versus Placebo in the Treatment of Trigger Finger: a Randomized Controlled Study
Brief Title: Extracorporeal Shock Wave in the Treatment of Trigger Finger
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N201810059
Record Dates: First submitted 2019-03-06; First posted 2019-04-26 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2018-11

CONDITIONS: Trigger Finger
Keywords: shock wave; trigger finger
MeSH Terms: conditions — Trigger Finger Disorder

STUDY DESIGN:
Intervention Model Description: Our pilot experiment on safety and effectiveness of Extracorporeal shock wave therapy (ESWT), we choose the two energy doses of ESWT for experiment:
  1. Low energy ESWT (1500 impulses and 0.006mJ/mm2, 3bar, once per week for 4 weeks)
  2. High energy ESWT (1500 impulses and 0.01mJ/mm2, 5.8bar, once per week for 4 weeks) In order to realize the effectiveness of ESWT on trigger finger, we will enroll a placebo group in which all participants will receive ESWT probe treatment with only vibration without transferring energy once per week for 4 weeks.
Who Masked: Participant, Outcomes Assessor
Masking Description: The patients will be randomized to each group. All participants are blinded to the treatment groups. All of the outcome will be followed by an assistant who is blinded to the allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low energy ESWT (Experimental): Low energy ESWT (using LITEMED"LM-ESWT-mini System with 1500 impulses and 0.006mJ/mm2, 3bar, once per week for 4 weeks)
  Interventions: Device: Low energy ESWT
- High energy ESWT (Experimental): High energy ESWT (using LITEMED"LM-ESWT-mini System with 1500 impulses and 0.01mJ/mm2, 5.8bar, once per week for 4 weeks)
  Interventions: Device: High energy ESWT
- Sham treatment (Sham Comparator): All participants will receive sham treatment using ESWT Probe with only vibration without transferring energy once per week for 4 weeks.
  Interventions: Device: Sham ESWT

INTERVENTIONS:
Device: Low energy ESWT — 1500 impulses and 0.006mJ/mm2, 3bar, once per week for 4 weeks
  Other Names: "LITEMED"LM-ESWT-mini System
  Arms: Low energy ESWT
Device: High energy ESWT — 1500 impulses and 0.01mJ/mm2, 5.8bar, once per week for 4 weeks
  Other Names: "LITEMED"LM-ESWT-mini System
  Arms: High energy ESWT
Device: Sham ESWT — sham treatment using ESWT Probe with only vibration without transferring energy once per week for 4 weeks
  Other Names: "LITEMED"LM-ESWT-mini System
  Arms: Sham treatment

SUMMARY:
Trigger finger (TF) is a condition that causes triggering, snapping, or locking on flexion of the involved finger, with a life- time risk between 2%-3% in the general population. A variety of treatments have been described, but the most effective treatment for this common disorder is still under debate. Recently, extracorporeal shock wave therapy(ESWT) has been advanced as a possible alternative to surgery for the treatment of musculoskeletal disorders in patients recalcitrant to traditional conservative treatment.

However, the effectiveness of ESWT on the treatment of TF is still in lack of evidence. The purpose of this study is to conduct a prospective randomized clinical trial to compare the efficacies of ESWT at two different energy flux density with placebo treatment for the management of TF. The investigators intended to enrolled 60 participants randomly allocated to three groups: low energy ESWT (1500 impulses and 0.006mJ/mm2, 3bar, once per week for 4 weeks), high energy ESWT (1500 impulses and 0.01mJ/mm2, 5.8bar, once per week for 4 weeks) or placebo treatment groups. The effectiveness of the treatment will be assessed using cure rates, a visual analogue scale, the frequency of triggering, the severity of triggering, the functional impact of triggering, and the Quick-Disabilities of the Arm, Shoulder, and Hand questionnaire (qDASH) at 1, 3, and 6 months after treatment. An intention-to-treat analysis will be used in this study. The investigators intend to determine the efficacy of ESWT in the treatment of TF and to find out the ideal energy set-up of ESWT for TF treatment.

DETAILED DESCRIPTION:
Trigger finger (TF) (also known as stenosing tenovaginitis) is characteristic of triggering, snapping, or locking on flexion of the involved metacarpophalangeal joint of finger, with incidence of 2%-3% in the general population and approximately 10% in diabetic patients. A variety of treatments have been described, including activity restriction, stretching exercise, splitting, non-steroid anti-inflammatory drugs, steroid injection, percutaneous or open release. However, none of the above-mentioned treatments is absolutely better than the others. The most effective treatment for this common disorder is still under debate.

Recently, extracorporeal shock wave therapy (ESWT) is getting popular as an alternative to surgery for the treatment of musculoskeletal disorders in patients recalcitrant to traditional conservative treatment. ESWT has been reported to effectively treat orthopedic disorders, such as plantar fasciitis, lateral epicondylitis of the elbow, calcific tendinopathies of the shoulder, and the non-union of long bone fractures. Biologically, ESWT is believed to result in a mechanosensitive feedback between the acoustic impulse and the stimulated cells, involving specific transduction pathways and gene expression. Furthermore, previous studies have shown that increased angiogenetic growth factors with ESWT are causally related to enhanced neovascularization and blood supply in the tendinopathy area of the tendon. ESWT can also induce the repair of the inflamed tissues by tissue regeneration and stimulates nitric oxide synthase, leading to suppression of ongoing inflammation in the soft tissues. However, there are still few clinical evidence on ESWT in treatment of TF in the literature.

One randomized control study reported the efficacy of ESWT in treatment of TF in 2016, and claimed that ESWT was as effective as steroid injection in treatment of TF. However, this clinical study was limited to the lack of control group with placebo treatment, since steroid injection for TF is reported to be with short-term effect and only effective in 57% of patients. Further evidence on the efficacy of ESWT in treatment of TF is needed to be clarified. In addition, the ideal energy set-up and protocol for ESWT are still left to be proven.

Considering the noninvasive advantage and potentially biological effect on the thickening of the flexor tendon and its sheath, the investigators hypothesize ESWT is effective on relieving the symptoms of TF. The purpose of this study is to conduct a prospective randomized clinical trial to compare the efficacies of ESWT at two different energy flux density with placebo treatment for the management of TF. The investigators intended to determine the efficacy of ESWT in the treatment of TF and to find out the ideal energy set-up of ESWT for TF treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Older than 20 years of age
2. Grade 2~3 trigger finger based on the Quinnell classification

Exclusion Criteria:

1. Previous treatment by physical therapy, local corticosteroid injection, or surgical release for trigger finger before the study
2. The presence of a musculoskeletal disease or previous nerve injuries at the upper extremities
3. Multiple trigger finger; local infection; malignancy; inflammatory arthritis; cardiac arrhythmia or cardiac pacemaker; and pregnancy.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-02-20 (Actual); Primary Completion 2019-11-22 (Estimated); Study Completion 2019-11-22 (Estimated)

PRIMARY OUTCOMES:
The efficacy of ESWT in the treatment of trigger finger | Baseline and Post-treatment 1, 3, 6 months
  Change from baseline the frequency of triggering, the severity of triggering and the functional impact of triggering at 1, 3, 6 months. We used a trigger finger assessment scale which included three 0- to 10- point subscales to determine the frequency, severity and functional impact of triggering to define the efficacy of treatment. In each subscale, the higher score means worse outcome. (Scale reference: Tarbhai K, Hannah S, von Schroeder HP: Trigger finger treatment: a comparison of 2 splint designs. J Hand Surg Am 2012, 37(2):243-249, 249.e241.)

SECONDARY OUTCOMES:
The change of Function Shoulder, and Hand questionnaire (qDASH) | Baseline and Post-treatment 1, 3, 6 months
  Functional evaluation utilizing the Quick-Disabilities of the Arm (q-DASH). The QuickDASH uses 11 items (scored 1-5) to measure physical function and symptoms in people with any or multiple musculoskeletal disorders of the upper limb. A higher score means worse disability.
The change of Pain | Baseline and Post-treatment 1, 3, 6 months
  evaluation utilizing Visual analogue scale (VAS). The visual analog scale (VAS) is an instrument regularly used to measure pain intensity based on a 0-10 cm. In the present trial, the researcher asked the patients: "Based on VAS, how much pain are you in/ experiencing?". The higher score means the more severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Pin Chen, M.D., Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University WanFang Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: starting 6 months after publication; ending 36 months after publication
Access Criteria: With whom: For investigators whose proposed use of the data has been approved by an independent committee
  For what type of analysis: For individual participants meta-analysis
  For what mechanism: To gain access, data requestor should sign a data access agreement. Data are available for 3 years at third party website.
URL: http://drive.google.com/drive/folders/16-F5ZqSK0srtbkXdshBX0L9Ur8WyaGMX?usp=sharing

REFERENCES:
- [Background] Koh S, Nakamura S, Hattori T, Hirata H. Trigger digits in diabetes: their incidence and characteristics. J Hand Surg Eur Vol. 2010 May;35(4):302-5. doi: 10.1177/1753193409341103. Epub 2009 Aug 17. PMID 19687073
- [Background] Strom L. Trigger finger in diabetes. J Med Soc N J. 1977 Nov;74(11):951-4. No abstract available. PMID 269967
- [Background] Amirfeyz R, McNinch R, Watts A, Rodrigues J, Davis TRC, Glassey N, Bullock J. Evidence-based management of adult trigger digits. J Hand Surg Eur Vol. 2017 Jun;42(5):473-480. doi: 10.1177/1753193416682917. Epub 2016 Dec 21. PMID 28488453
- [Background] Romeo P, Lavanga V, Pagani D, Sansone V. Extracorporeal shock wave therapy in musculoskeletal disorders: a review. Med Princ Pract. 2014;23(1):7-13. doi: 10.1159/000355472. Epub 2013 Nov 5. PMID 24217134
- [Background] Yin M, Chen N, Huang Q, Marla AS, Ma J, Ye J, Mo W. New and Accurate Predictive Model for the Efficacy of Extracorporeal Shock Wave Therapy in Managing Patients With Chronic Plantar Fasciitis. Arch Phys Med Rehabil. 2017 Dec;98(12):2371-2377. doi: 10.1016/j.apmr.2017.05.016. Epub 2017 Jun 17. PMID 28634056
- [Background] Yang TH, Huang YC, Lau YC, Wang LY. Efficacy of Radial Extracorporeal Shock Wave Therapy on Lateral Epicondylosis, and Changes in the Common Extensor Tendon Stiffness with Pretherapy and Posttherapy in Real-Time Sonoelastography: A Randomized Controlled Study. Am J Phys Med Rehabil. 2017 Feb;96(2):93-100. doi: 10.1097/PHM.0000000000000547. PMID 27323324
- [Background] Arirachakaran A, Boonard M, Yamaphai S, Prommahachai A, Kesprayura S, Kongtharvonskul J. Extracorporeal shock wave therapy, ultrasound-guided percutaneous lavage, corticosteroid injection and combined treatment for the treatment of rotator cuff calcific tendinopathy: a network meta-analysis of RCTs. Eur J Orthop Surg Traumatol. 2017 Apr;27(3):381-390. doi: 10.1007/s00590-016-1839-y. Epub 2016 Aug 23. PMID 27554465
- [Background] Alkhawashki HM. Shock wave therapy of fracture nonunion. Injury. 2015 Nov;46(11):2248-52. doi: 10.1016/j.injury.2015.06.035. Epub 2015 Jul 3. PMID 26323379
- [Background] Cacchio A, Giordano L, Colafarina O, Rompe JD, Tavernese E, Ioppolo F, Flamini S, Spacca G, Santilli V. Extracorporeal shock-wave therapy compared with surgery for hypertrophic long-bone nonunions. J Bone Joint Surg Am. 2009 Nov;91(11):2589-97. doi: 10.2106/JBJS.H.00841. PMID 19884432
- [Background] Hsu RW, Hsu WH, Tai CL, Lee KF. Effect of shock-wave therapy on patellar tendinopathy in a rabbit model. J Orthop Res. 2004 Jan;22(1):221-7. doi: 10.1016/S0736-0266(03)00138-4. PMID 14656684
- [Background] Orhan Z, Ozturan K, Guven A, Cam K. The effect of extracorporeal shock waves on a rat model of injury to tendo Achillis. A histological and biomechanical study. J Bone Joint Surg Br. 2004 May;86(4):613-8. PMID 15174564
- [Background] Seok H, Kim SH. The effectiveness of extracorporeal shock wave therapy vs. local steroid injection for management of carpal tunnel syndrome: a randomized controlled trial. Am J Phys Med Rehabil. 2013 Apr;92(4):327-34. doi: 10.1097/PHM.0b013e31826edc7b. PMID 23044704
- [Background] Yildirim P, Gultekin A, Yildirim A, Karahan AY, Tok F. Extracorporeal shock wave therapy versus corticosteroid injection in the treatment of trigger finger: a randomized controlled study. J Hand Surg Eur Vol. 2016 Nov;41(9):977-983. doi: 10.1177/1753193415622733. Epub 2016 Sep 28. PMID 26763271
- [Background] Fleisch SB, Spindler KP, Lee DH. Corticosteroid injections in the treatment of trigger finger: a level I and II systematic review. J Am Acad Orthop Surg. 2007 Mar;15(3):166-71. doi: 10.5435/00124635-200703000-00006. PMID 17341673
- [Derived] Chen YP, Lin CY, Kuo YJ, Lee OK. Extracorporeal Shockwave Therapy in the Treatment of Trigger Finger: A Randomized Controlled Study. Arch Phys Med Rehabil. 2021 Nov;102(11):2083-2090.e1. doi: 10.1016/j.apmr.2021.04.015. Epub 2021 May 21. PMID 34029555